CLINICAL TRIAL: NCT02208466
Title: Effects of Contralesional Repetitive Magnetic Stimulation Combined With Fluoxetine on Motor Recovery in Acute Stroke Patients
Brief Title: Effects rTMS Combined With Fluoxetine on Motor Recovery in Stroke Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P001046
Record Dates: First submitted 2014-07-28; First posted 2014-08-05 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Motor Function
Keywords: repetitive transcranial magnetic stimulation; rTMS; TMS; fluoxetine
MeSH Terms: conditions — Stroke | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active rTMS/active fluoxetine (Experimental): Subjects in this arm will undergo 10 daily sessions over 15 days of active low-frequency rTMS with each session lasting 20 minutes. This will be followed by 8 weekly sessions of active low-frequency rTMS with each session lasting 20 minutes. Additionally, during this time beginning with enrollment, subjects will also be taking 20mg of active fluoxetine by mouth daily.
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS); Drug: Fluoxetine
- Sham rTMS/active fluoxetine (Experimental): Subjects in this arm will undergo 10 daily sessions over 15 days of sham low-frequency rTMS with each session lasting 20 minutes. This will be followed by 8 weekly sessions of sham low-frequency rTMS with each session lasting 20 minutes. Additionally, during this time beginning with enrollment, subjects will also be taking 20mg of active fluoxetine by mouth daily.
  Interventions: Drug: Fluoxetine; Device: Sham repetitive transcranial magnetic stimulation (rTMS)
- Sham rTMS/placebo fluoxetine (Experimental): Subjects in this arm will undergo 10 daily sessions over 15 days of sham low-frequency rTMS with each session lasting 20 minutes. This will be followed by 8 weekly sessions of sham low-frequency rTMS with each session lasting 20 minutes. Additionally, during this time beginning with enrollment, subjects will also be taking 20mg of placebo fluoxetine by mouth daily.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation (rTMS); Drug: Placebo Fluoxetine

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS) — Subjects will undergo active low-frequency rTMS (1Hz continuous). Each session will last 20 minutes and will be conducted at 100% of the motor threshold.
  Other Names: magnetic stimulation, Magstim
  Arms: Active rTMS/active fluoxetine
Drug: Fluoxetine — Subjects will receive active fluoxetine (20mg) and take orally consecutively for 90 days.
  Other Names: Prozac, Sarafem, Ladose, Fontex
  Arms: Active rTMS/active fluoxetine; Sham rTMS/active fluoxetine
Device: Sham repetitive transcranial magnetic stimulation (rTMS) — Subjects will undergo sham low-frequency rTMS (using sham coil). This session will last 20 minutes, just as the active session would, however, no magnetic pulses will be delivered.
  Other Names: Magstim, magnetic stimulation
  Arms: Sham rTMS/active fluoxetine; Sham rTMS/placebo fluoxetine
Drug: Placebo Fluoxetine — Subject will receive placebo fluoxetine (sugar pills) and will take orally consecutively for 90 days.
  Other Names: Prozac, Sarafem, Ladose, Fontex
  Arms: Sham rTMS/placebo fluoxetine

SUMMARY:
In this study investigator's aim to assess the effect of a type of non-invasive brain stimulation technique called repetitive transcranial magnetic stimulation (rTMS) in conjunction with fluoxetine on motor recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic infarction within the past 2 years post event that has caused hemiparesis or hemiplegia, as self-reported and/or confirmed by medical record.
* Older than 18 years old.
* Upper extremity weakness defined as a score of >11 and ≤56 on the arm motor Fugl-Mayer motor scale.
* Minimal pre-stroke disability defined as a score of <3 in the Modified Rankin Scale.
* Subjects need to be able to follow directions and participate in 2 hours of testing with short breaks.
* Subjects need to be able to provide informed consent.

Exclusion Criteria:

* Any substantial decrease in alertness, language reception, or attention that might interfere with understanding instruction for motor testing
* Excessive pain in any joint of the paretic extremity (not applicable to severe stroke subjects), as self reported
* Contraindications to single pulse TMS (will be used to measure cortical excitability) such as: history of seizures, unexplained loss of consciousness, any metal implants in the head, frequent or severe headaches or neck pain, any other electronic implanted medical devices such as pacemakers, defibrillators, or implant medication pump.
* Patients who have taken fluoxetine in the past 5 weeks.
* Patients taking any other SSRI at the time of enrollment or in the previous month.
* Patients taking any other medication likely to have adverse interaction with SSRIs (all the medications the patient is taking will be carefully reviewed, as noted below in "Monitoring of important drug interactions").
* Active depression on admission to SRH defined by a score of 24 or higher in the Hamilton Depression Rating Scale (HAM-D)
* Concurrent medical condition likely to worsen patient's functional status in the next 6 months such as: cancer, terminal heart, kidney or liver disease, as self-reported and/or confirmed by medical record.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-09; Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PhD MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Derived] Bonin Pinto C, Morales-Quezada L, de Toledo Piza PV, Zeng D, Saleh Velez FG, Ferreira IS, Lucena PH, Duarte D, Lopes F, El-Hagrassy MM, Rizzo LV, Camargo EC, Lin DJ, Mazwi N, Wang QM, Black-Schaffer R, Fregni F. Combining Fluoxetine and rTMS in Poststroke Motor Recovery: A Placebo-Controlled Double-Blind Randomized Phase 2 Clinical Trial. Neurorehabil Neural Repair. 2019 Aug;33(8):643-655. doi: 10.1177/1545968319860483. Epub 2019 Jul 9. PMID 31286828

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that from the 44 subjects enrolled, only 27 started (were randomized) as 17 subjects screened out during confirmation of eligibility after signing the consent form (some of the criteria could only be checked after consent).
Period: Overall Study
Arm/Group | Active rTMS/Active Fluoxetine | Sham rTMS/Active Fluoxetine | Sham rTMS/Placebo Fluoxetine
Started | 9 | 10 | 8
Completed | 9 | 10 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS/Active Fluoxetine | Sham rTMS/Active Fluoxetine | Sham rTMS/Placebo Fluoxetine | Total
Number analyzed (Participants) | 9 | 10 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.22 (9.39) | 50.5 (16.57) | 57.38 (9.96) | 55.03 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 2 | 11
  Male | 5 | 5 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 5
  White | 8 | 9 | 5 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Motor Function (Jebsen-Taylor Task)
Description: Jebsen Taylor Hand Function Test: measures hand function in real-life activities, by evaluating the time required to perform 7 different tasks. We used the non-constrained hand for the assessments. The sum of the different tasks was used for the analysis.
  Calculation details: value at 9 months minus value at baseline, change in seconds (adjusted mean difference).
Time Frame: baseline and 90 days
Population: Performed by a rater blinded to rTMS and pharmacotherapy performed all assessments
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Active rTMS/Active Fluoxetine | Sham rTMS/Active Fluoxetine | Sham rTMS/Placebo Fluoxetine
Number analyzed (Participants) | 9 | 10 | 8
seconds | -214.33 [-289.32 to -139.35] | -50.16 [-110.56 to -10.24] | -117.98 [-197.39 to -38.58]

2. Primary Outcome: Changes in Fugl-Meyer Assessment (FMA) Scale
Description: The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation, and joint functioning in patients with post-stroke hemiplegia. We used the upper limb motor function subscale: minimum values= 0 ; maximum values= 66. Higher scores mean a better outcome. Changes from baseline to 90 days (value at 90 days minus value at baseline).
Time Frame: baseline and 90 days
Population: Performed by a rater blinded to rTMS and pharmacotherapy performed all assessments
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active rTMS/Active Fluoxetine | Sham rTMS/Active Fluoxetine | Sham rTMS/Placebo Fluoxetine
Number analyzed (Participants) | 9 | 10 | 8
units on a scale | 10.10 [4.06 to 16.14] | 6.73 [1.28 to 12.17] | 15.55 [9.16 to 21.95]

3. Secondary Outcome: Changes in Cortical Excitability Measures
Description: We will measure cortical excitability using single-pulsed transcranial magnetic stimulation (TMS) before and after stimulation at three different time-points. Changes from baseline to 90 days (value at 90 days minus value at baseline).
Time Frame: Baseline and 90 days
Population: Performed by a rater blinded to rTMS and pharmacotherapy performed all assessments
Measure: Mean (95% Confidence Interval); unit: motor evoked potential (mV)
Arm/Group | Active rTMS/Active Fluoxetine | Sham rTMS/Active Fluoxetine | Sham rTMS/Placebo Fluoxetine
Number analyzed (Participants) | 9 | 10 | 8
motor evoked potential (mV) | -0.05 [-0.34 to 0.08] | -0.12 [-0.33 to 0.43] | 0.33 [0.07 to 1.16]

ADVERSE EVENTS:
Time Frame: 3 months
Description: adverse effects were collected with a questionnaire for adverse effects
Arm/Group | Active rTMS/Active Fluoxetine | Sham rTMS/Active Fluoxetine | Sham rTMS/Placebo Fluoxetine
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 2/9 | 0/10 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS/Active Fluoxetine (N=9) | Sham rTMS/Active Fluoxetine (N=10) | Sham rTMS/Placebo Fluoxetine (N=8)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT02208466/Prot_SAP_000.pdf